CLINICAL TRIAL: NCT00020657
Title: Treatment of Delayed Nausea: What Works Best?
Brief Title: Comparison of Antiemetic Drugs in Preventing Delayed Nausea After Chemotherapy in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, University of Rochester NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000068694; URCC-U3901; NCI-P01-0180
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Nausea; Vomiting | interventions — dolasetron; Granisetron; Ondansetron; Prochlorperazine

INTERVENTIONS:
Drug: dolasetron mesylate
Drug: granisetron hydrochloride
Drug: ondansetron
Drug: prochlorperazine
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Antiemetic drugs may help to reduce or prevent nausea and vomiting in patients being treated with chemotherapy.

PURPOSE: This randomized phase III trial is comparing how well different antiemetic drugs work in preventing delayed nausea after chemotherapy in patients who have cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of a 5 hydroxytryptamine 3 (5-HT3) receptor antagonist antiemetic vs prochlorperazine in controlling delayed nausea after chemotherapy in patients with chemotherapy-naive cancer.
* Compare the effectiveness of prochlorperazine administered on a preventive vs as needed basis in controlling delayed nausea after chemotherapy in these patients.
* Compare the quality of life of patients treated with a 5-HT3 receptor antagonist antiemetic vs prochlorperazine.
* Compare the quality of life of patients treated with prochlorperazine administered on a preventive vs as needed basis.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center.

Patients receive their scheduled chemotherapy regimen containing doxorubicin and their scheduled oral 5 hydroxytryptamine 3 receptor antagonist antiemetic (ondansetron, granisetron, tropisetron, or dolasetron mesylate) combined with dexamethasone on day 1.

Patients are then randomized to 1 of 3 antiemetic arms.

* Arm I: Patients receive oral prochlorperazine every 8 hours on days 2 and 3.
* Arm II: Patients receive oral ondansetron every 12 hours, oral granisetron every 12 hours, or oral dolasetron mesylate either once a day or every 12 hours on days 2 and 3.
* Arm III: Patients receive oral prochlorperazine as needed, up to 4 times per day, on days 2 and 3.

Quality of life is assessed at baseline and on day 4.

PROJECTED ACCRUAL: A total of 670 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer for which a chemotherapy regimen containing doxorubicin (with adjuvant, neoadjuvant, curative, or palliative intent) is scheduled
* Scheduled chemotherapy regimen must not include any of the following:

  * Multiple doses of doxorubicin, dacarbazine, hexamethylmelamine, nitrosoureas, or streptozocin
  * Doxorubicin HydroCloride liposome or cisplatin
* Scheduled chemotherapy regimen may contain agents, other than those listed above, administered orally, IV, or IV continuously on 1 or multiple days
* Must be scheduled to receive a 5 hydroxytryptamine 3 (5-HT3) receptor antagonist antiemetic (ondansetron, granisetron, tropisetron, or dolasetron mesylate) with dexamethasone concurrently with doxorubicin
* No clinical evidence of an impending bowel obstruction
* No symptomatic brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent interferon

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* Concurrent rescue medications (as appropriate) for control of symptoms caused by cancer or its treatment allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Morrow, PhD, MS, Study Chair — James P. Wilmot Cancer Center
Locations (15):
- United States (15):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - CCOP - North Shore University Hospital, Manhasset, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Hickok JT, Roscoe JA, Morrow GR, Bole CW, Zhao H, Hoelzer KL, Dakhil SR, Moore T, Fitch TR. 5-Hydroxytryptamine-receptor antagonists versus prochlorperazine for control of delayed nausea caused by doxorubicin: a URCC CCOP randomised controlled trial. Lancet Oncol. 2005 Oct;6(10):765-72. doi: 10.1016/S1470-2045(05)70325-9. Epub 2005 Sep 13. PMID 16198982